CLINICAL TRIAL: NCT00981279
Title: Profile of HIV Seropositive Patients on Antiretroviral Therapy at the Clinical Hospital of the Federal University of Goiás
Brief Title: Profile of HIV Seropositive Patients
Acronym: PHSP
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Caroline Nayanna Rodrigues Santos, Universidade Federal de Goiás
Other Study IDs: 129/2009; CONEP- 129/2009
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infection; HIV Infections
Keywords: Health Profile; AIDS; Health Promotion; HIV; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV seroposite patients: Seroposite HIV patients that take their treatment at the Clinical Hospital of The Federal University of Goias, and have their records in the hospital.

SUMMARY:
The aim of this study was to delineate the epidemiological profile of HIV seropositive patients on antiretroviral therapy at the Clinical Hospital of the Federal University of Goiás.

DETAILED DESCRIPTION:
Objective: To delineate the epidemiological profile of HIV seropositive patients on antiretroviral therapy at the Clinical Hospital of the Federal University of Goiás.

Methods: The present study is documental and analitical descriptive and it was conducted at the Clinical Hospital of the Federal University of Goiás, trough data collection of 222 records of individuals in drug therapy. Data were collected regarding the personal aspects, aspects related to the infection and information about the most used therapeutic.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients that had data in the hospital
* All with the diagnose of HIV
* Using antiretroviral drugs

Exclusion Criteria:

* Incompleted records
* Patients who didn't take their medicines regularly.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample, with HIV, in drug therapy in the Clinical Hospital of UFG.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Data regarding the personal aspects, aspects related to the infection and information about the most used therapeutic. | Since the start of the drug therapy ( means of 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline N Rodrigues, Graduated, Principal Investigator — UFG
Locations (1):
- Federal University of Goias, Goiânia, Goiás, Brazil

REFERENCES:
- See also: Information about epidemiological datas of HIV patients in Goiás, Brazil — http://www.saude.go.gov.br/index.php?idMateria=16409